CLINICAL TRIAL: NCT00812916
Title: EXPRESSO - European Carto® XP REgistry for Validating Specialized CFAE SOftware
Brief Title: European Carto® XP REgistry for Validating Specialized CFAE SOftware
Acronym: EXPRESSO
Status: Completed | Type: Observational
Sponsor: Biosense Webster EMEA (Industry)
Responsible Party: Sponsor
Organization: Biosense Webster, Inc. (Industry)
Other Study IDs: EXPRESSO
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
Keywords: Persistent or longstanding persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RF ablation: RF Ablation using specialized CFAE software
  Interventions: Procedure: RF ablation, using specialized CFAE software

INTERVENTIONS:
Procedure: RF ablation, using specialized CFAE software — RF ablation

SUMMARY:
The purpose of this prospective observational study (registry) is to determine the acute success rate of a complex fractionated atrial electrogram (CFAE) guided ablation procedure using a dedicated software and to determine the functionality and performance of the CFAE software in patients with a type of persistent atrial fibrillation (AF) in routine clinical practice.

DETAILED DESCRIPTION:
This was a prospective, multi-center, observational registry study evaluating CARTO® XP CFAE Software (CFAE Software) in subjects with chronic AF requiring CFAE-guided RFCA. Use of the CARTO® 3 System (including CFAE Software) was also allowed. The primary efficacy endpoint was the acute success rate of CFAE-guided radiofrequency catheter ablation (RFCA) using the CFAE Software. Acute success is defined as the subject achieving sinus rhythm at the end of the procedure without electrical or pharmaceutical cardioversion. Secondary endpoints consisted of measures of efficacy (example, performance of the CFAE Software) and of safety (example, number of procedure-related adverse events).

ELIGIBILITY:
Inclusion Criteria:

* Persistent or longstanding persistent AF

Exclusion Criteria:

* Previously underwent RF ablation for AF and patients with paroxysmal AF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with persistent or longstanding persistent atrial fibrillation (AF), needing radiofrequency (RF) ablation
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Albenque, MD, Principal Investigator — Clinique Pasteur - Unité de Cardiologie interventionnelle; Agustin Bortone, MD, Principal Investigator — Hôpital Les Franciscaines Service Rhythmologie,; André Pisapia, MD, Principal Investigator — Hôpital Saint Joseph; Franck Raczka, MD, Principal Investigator — CHU Arnaud de Villeneuve; Csaba Földesi, MD, Principal Investigator — Gottsegen György Országos Kardiológiai Intézet; Armin Luik, MD, Principal Investigator — Städtisches Klinikum Karlsruhe; Boris Schmidt, MD, Principal Investigator — Asklepios Klinik St. Georg; Ahmed Abdelaal, MD, Principal Investigator — Central Hospital, Nancy, France; Gilles-Sélim Lande-Abbey, MD, Principal Investigator — Hôpital Laënnec - CHU de Nantes; Bruno Cauchemez, MD, Principal Investigator — Clinique Ambroise Paré; Nicolas Lellouche, MD, Principal Investigator — Henri Mondor University Hospital; Fabrice Extramiana, MD, Principal Investigator — Hôpital Lariboisière Service de Rhytmologie; Julien Seitz, MD, Principal Investigator — Hôpital Privé Jacques Cartier Service de Rhytmologie
Locations (13):
- France (10):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Saint Joseph, Marseille
  - Hôpital Privé Jacques Cartier Service de Rhytmologie, Massy
  - CHU Arnaud de Villeneuve, Montpellier
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Hôpital Les Franciscaines Service Rhythmologie, Nîmes
  - Hôpital Lariboisière Service de Rhytmologie, Paris
  - Hôpital Laënnec - CHU de Nantes, Saint-Herblain
  - Clinique Pasteur - Unité de Cardiologie interventionnelle, Toulouse
  - CHU de Nancy, Vandœuvre-lès-Nancy
- Germany (2):
  - Asklepios Klinik St. Georg, Hamburg
  - Städtisches Klinikum Karlsruhe, Karlsruhe
- Gottsegen György Országos Kardiológiai Intézet, Budapest, Hungary

RESULTS

PARTICIPANT FLOW:
Groups:
- Number of Patients: Radiofrequency (RF) Ablation using specialized complex fractionated atrial electrogram (CFAE) software
Period: Overall Study
Arm/Group | Number of Patients
Started | 206 (206 enrolled (consented))
Data Available | 205
CFAE - Guided Ablation | 203
Completed | 203
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Enrolled patients
Groups:
- Radiofrequency (RF) Ablation: RF Ablation using specialized complex fractionated atrial electrogram (CFAE) software
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 206
Age, Customized [Number; unit: participants] — Age and gender were not collected for this trial.
  participants
    Not Collected | 206
Sex/Gender, Customized [Number; unit: participants] — Age and gender were not collected for this trial.
  participants
    Not Collected | 206

OUTCOME MEASURES:

1. Primary Outcome: Acute Success
Description: Sinus rhythm achieved at end of ablation procedure without electrical or pharmaceutical cardioversion
Time Frame: End of procedure
Population: Patients with CFAE-guided RF catheter ablation
Measure: Number (95% Confidence Interval); unit: percentage achieving success
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 203
percentage achieving success | 48.8 [41.7 to 55.9]

2. Secondary Outcome: Total Ablation Time
Description: Total time of ablation with exception of 10 outliers with >180 minutes of total ablation time reported
Time Frame: Procedural
Population: Safety population with ablation time reported
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 188
minutes | 61.4 (42.0)

3. Secondary Outcome: Total Complex Fractionated Atrial Electrogram (CFAE) Mapping Time
Description: Total of left and right atrium CFAE mapping times with exception of 9 outliers reporting total CFAE mapping time of >120 minutes
Time Frame: Procedural
Population: Safety population with mapping time reported
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Radiofrequency (RF) Ablation: RF Ablation using specialized CFAE software
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 193
minutes | 27.7 (15.4)

4. Secondary Outcome: Total Radiofrequency (RF) Duration
Description: Total duration of all radiofrequency applications with exception of 12 outliers recording >150 minutes.
Time Frame: Procedural
Population: Safety population with RF data reported
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- RF Ablation: RF Ablation using specialized complex fractionated atrial electrogram (CFAE) software
Arm/Group | RF Ablation
Number analyzed (Participants) | 173
minutes | 76.2 (24.8)

5. Secondary Outcome: Total Fluoroscopy Time
Description: Mean total fluoroscopy time
Time Frame: Procedural
Population: Safety population with fluoroscopy time reported
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 192
minutes | 43.3 (28.6)

6. Secondary Outcome: Total Number of Ablated Complex Fractionated Atrial Electrogram (CFAE) Discrete Points
Description: Does not include 2 outliers with >300 CFAE discrete points. Based on the user-defined definition of a CFAE complex, the system identifies the number of intervals between adjacent CFAE complexes and the cycle length of these intervals. This makes it possible to estimate the number of CFAE complexes within certain amplitude and duration values. A CFAE complex is defined by the system based on the intervals between the peaks. Therefore, clinically, the CFAE software includes an algorithm that enables detection of CFAE complexes. The automatic detection and distribution of CFAE signals is taking place during a 2.5 second intra-cardiac ECG recording. When the CFAE areas are completely eliminated, but the arrhythmia continues as organized atrial flutter or atrial tachycardia, the atrial tachy-arrhythmias may be mapped and ablated upon discretion of the investigator. Analyses occur post-procedure.
Time Frame: Procedural
Population: Safety population with non-outlier endpoint reported
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 193
points | 33.5 (43.1)

ADVERSE EVENTS:
Time Frame: Peri-procedural, up to duration of study
Description: Procedure and/or device related
Arm/Group | Radiofrequency (RF) Ablation
Serious Adverse Events (participants affected / at risk) | 13/205
Other Adverse Events (participants affected / at risk) | 3/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiofrequency (RF) Ablation (N=205)
Tamponade (Cardiac disorders) | 1
Sheath retained in femoral vein (Injury, poisoning and procedural complications) | 1
Pericardial effusion (Cardiac disorders) | 6
Epicardial effusion (Cardiac disorders) | 1
Hematoma (Injury, poisoning and procedural complications) | 2
Phrenic nerve injury (Injury, poisoning and procedural complications) | 1
Pleural tamponade (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiofrequency (RF) Ablation (N=205)
Pericardial effusion (Cardiac disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.